CLINICAL TRIAL: NCT06607744
Title: The Comparative Pilot Bioavailability Study of a Generic Test Formulation of Selegiline TDS 6 mg/24 Hours Against the Comparator EMSAM® 6 mg/24 Hours in Healthy Adult Subjects
Brief Title: Determine the Bioavailability of Selegiline TDS 6mg/24 Hours vs EMSAM in Healthy Subjects
Acronym: TDS
Status: Recruiting | Type: Observational
Sponsor: Corium Innovations, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SE101
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: MDD
Keywords: Selegiline TDS; Bioavailability; Pharmacokinetic
MeSH Terms: interventions — Selegiline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Days
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group1: Selegiline TDS of test formulation (6mg/24 hours): Group1: 1 x Selegiline TDS 6 mg/24 hours manufactured by Corium Innovations, Inc., worn over 24 hours on cleaned upper left or right arm approximately from 8 AM following the randomisation schedule.
  Interventions: Drug: Pharmacokinetic profiles of Selegiline TDS and EMSAM
- Group2: EMSAM TDS (6 mg/24 hours): 1 x EMSAM® TDS 6 mg/24 hours manufactured by Somerset Pharmaceuticals, Inc., worn over 24 hours on cleaned upper left or right arm approximately from 8 AM following the randomisation schedule.
  Interventions: Drug: Pharmacokinetic profiles of Selegiline TDS and EMSAM

INTERVENTIONS:
Drug: Pharmacokinetic profiles of Selegiline TDS and EMSAM — Selegiline concentrations will be measured in blood plasma using a validated liquid chromatography tandem mass spectrometry method from Selegiline TDS (test formulation 6mg/24 hours) and EMSAM (6mg/24 hours). The analytical laboratory will be blinded as to samples which are the test and reference products.
  Other Names: Systemic and local tolerability

SUMMARY:
The goal of this clinical study is to obtain the bioavailability of the test patch of a generic formulation of Selegiline TDS 6mg/24 hours by Corium Innovations against the comparator (EMSAM), and the systemic and local safety and tolerability will be also observed and evaluated.

DETAILED DESCRIPTION:
This is a pilot, single-dose, single-centre, open-label, randomised, 2-way crossover study (2 treatments, 2 periods and 2 sequences) of a generic test formulation of Selegiline TDS 6 mg/24 hours with the comparator EMSAM® TDS 6 mg/24 hours, with at least 14 days washout period, recruiting around 12 healthy male and female subjects.

For each study period, subjects will be admitted and confined in the clinical study site the night before the study day from at least 10 hours before dosing and they will be discharged once all PK, safety and tolerability are completed at 36 hours after dosing. Subjects will be required to return for subsequent PK, safety and tolerability at 48-, 72- and 96-hours post-dosing. The clinic will follow up by telephone 7 ± 3 days after completion of the study.

Pharmacokinetic Blood Sampling:

PK blood samples will be collected before dosing and at 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 24, 30, 36, 48, 72, 96 hours after dosing.

Pharmacokinetics:

PK parameters include AUC0-t, AUC0-∞, Cmax, tmax, t½, tlag (if applicable), λz, and Mean residence time (MRT) will be evaluated for Selegiline.

Safety:

Safety will be assessed on all subjects who participate in the study from the beginning to the end. Adverse events (AEs), abnormal vital signs, abnormal ECG results, abnormal physical examination findings and abnormal clinical laboratory test results will be reviewed on a subject-to-subject basis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age between 18 to 55 years old with adequate contraception but without taking oral contraceptives.
2. Subject body weight ≤ 120 kg, with a BMI within 18-30 kg/m².
3. Subject is able to complete the clinical study including the follow-up.
4. Subject is capable of providing written informed consent.
5. Subjects are able and willing to follow the requirements of the study and wearing patches.

Exclusion Criteria:

1. Breastfeeding female.
2. Pregnancy test positive female.
3. At rest systolic blood pressure outside 90-140 mmHg or diastolic blood pressure outside 50- 90 mmHg or orthostatic hypotension.
4. At rest sinus bradycardia defined as symptomatic heart rate < 50 bpm, or asymptomatic heart rate < 45 bpm; and sinus tachycardia defined as heart rate > 100 bpm.
5. Clinically significant ECG abnormalities (PQ interval > 0.2 s, Duration of the QRS complex > 0.1 s, AV block).
6. QTc > 450 ms for male and > 460 ms for female.
7. A history of allergies, or any significant adverse reactions, to any medications, unless the clinician considers that they are not clinically significant.
8. Clinically significant medical history of eyes, ears, nose, throat, respiratory, cardiovascular, gastrointestinal, genitourinary, neurological, haematopoietic, lymphatic, endocrine, metabolic, dermatological, musculoskeletal, psychological, family history or surgical history.
9. Family history of sudden cardiac death or pheochromocytoma.
10. Clinically significant physical examination finding or psychiatric unstable conditions or psychiatric illness requiring treatment.
11. Clinically significant laboratory abnormalities.
12. Haemoglobin < 12.0 g/dL for male and < 11.0 g/dL for female at screening.
13. Total bilirubin > 1.25 x upper limit of normal, ALT/AST > 1.5 x upper limit of normal.
14. Hepatitis B, Hepatitis C or HIV positive.
15. Urine DOA test positive.
16. Breath alcohol test positive.
17. Any smoker with tobacco or electronic tobacco products.
18. A history of drug or substance abuse, including alcohol (≥ 14 units per week) within 6 months before consent taking (1 unit of alcohol equals approximately ½ pint [285 mL] of beer, 1 glass [125 mL] of wine, or 1 shot [25 mL] of spirit).
19. Taking selective serotonin reuptake inhibitors (SSRI), serotonin and norepinephrine reuptake inhibitors (SNRI) or cough or cold medicine (e.g., dextromethorphan, pseudoephedrine) or using carbamazepine or oxcarbazepine, or using meperidine and analgesic agents such as tramadol, methadone, and propoxyphene, or using sympathomimetic agents.
20. Unable to refrain from taking any medications (including herbal remedies) within 7 days before dosing, with the exception of birth control medications and other medications deemed acceptable by the Investigator.
21. Clinically significant illness or injury or hospitalisation for any reason within 28 days before consent taking.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological sex
Study Population: Local subjects participate in the Hospital Ampang, Malaysia
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Plasma Pharmacokinetic-AUC 0-t | 22 days
  The area under the plasma concentration-time curve from time 0 to the last measurable concentration is calculated by the linear/log trapezoidal method where the liner trapezoidal method is applied up to Tmax and the log trapezoidal method is used after Tmax.
Plasma Pharmacokinetic-AUC 0-∞ | 22 days
  The area under the plasma concentration-time curve from time 0 to infinity is calculated as the sum of AUC0-t and Ct/Kel, where Ct is the last measurable concentration.
Plasma Pharmacokinetic-Cmax | 22 days
  The maximum plasma concentration following drug administration
Plasma Pharmacokinetic-Tmax | 22 days
  The time to achieve maximum plasma concentration is determined directly from the individual plasma concentration-time curves
Plasma Pharmacokinetic-T1/2 | 22 days
  The terminal elimination half-life is calculated as 0.693/Kel
Plasma Pharmacokinetic-Tlag | 22 days
  The time prior to achieving the first measurable plasma concentration (if applicable)
Plasma Pharmacokinetic-MTR | 22 days
  The mean residence time
Plasma Pharmacokinetic-λz (Lambda z) | 22 days
  Individual estimate of the terminal elimination rate constant, calculated using log-linear regression of the terminal portions of the plasma concentration-versus-time curves

SECONDARY OUTCOMES:
Safety-Topic Skin Irritation | 22 days
  Each application site will receive a separate dermal response score and other effect score. Dermal response scores require that at least 25% or more of the patch area demonstrate an observable response. The percentage of the patch area demonstrating an observable response will also be recorded. "Strong" reaction to the transdermal patch is defined as a dermal response score of 3-7 or any dermal response score combined with other effect score of 4 or greater.

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Hospital Ampang, Pandan Mewah, Ampang
  - Sarawak General Hospital, Samoran, Sarawak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Approved Drugs — https://www.accessdata.fda.gov/scripts/cder/daf/index.cfm?event=overview.process&ApplNo=021336